CLINICAL TRIAL: NCT03169114
Title: Raja Isteri Pengiran Anak Saleha Appendicitis Treatment Without Operation - Antibiotic Non-operative Management Strategy Versus Surgery Management Strategy, a Non-Inferiority Randomised Controlled Trial.
Brief Title: Raja Isteri Pengiran Anak Saleha Appendicitis Treatment Without Operation
Acronym: RIPASA-TWO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment and terminated during COVID-19 pandemic
Sponsor: Raja Isteri Pengiran Anak Saleha Hospital (Other Government)
Responsible Party: Principal Investigator, William Chong Chee Fui, Consultant Surgeon, Raja Isteri Pengiran Anak Saleha Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ripas
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Appendicitis; Surgery
Keywords: Appendicitis; Surgery; Antibiotic therapy; RIPASA Score
MeSH Terms: conditions — Appendicitis | interventions — Amikacin; Appendectomy

STUDY DESIGN:
Intervention Model Description: Non-Inferiority Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors - Histopathologists will be masked in terms of allocation of the study participants, when reporting histology specimen of appendix removed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amikacin injection (Active Comparator): Antibiotic Non-Operative Management Strategy
  Interventions: Drug: Amikacin Injection
- Appendicectomy (Active Comparator): Surgery Management Strategy
  Interventions: Procedure: Appendicectomy

INTERVENTIONS:
Drug: Amikacin Injection — Participants allocated to Antibiotic Non-operative Management Strategy will be given intravenous Amikacin 15mg/kg/day divided over 3 doses for first 48 hours and followed by oral ciprofloxacin 500mg bd for 7 days
  Other Names: Amikin
  Arms: Amikacin injection
Procedure: Appendicectomy — Patients allocated to Surgery Management Strategy will undergo appendicectomy
  Other Names: Appendectomy
  Arms: Appendicectomy

SUMMARY:
The RIPASA score is a Clinical Prediction Rule (CPR) for the diagnosis of acute appendicitis. Since its inception in 2009, the RIPASA score has been validated in various population in healthcare institutions around the world and reported significantly higher sensitivity and specificity when compared to Alvarado score. RIPASA score ranges from 3 to 16.5 with those having a score of less than 7 having a low probability of acute appendicitis and those with a score of 7.5 having a high probability of acute appendicitis.

There has been a trend in the past decade on non-operative management of early-uncomplicated acute appendicitis (EuAA) with antibiotic therapy. This antibiotic non-operative management strategy (AMS) has been reported to work in children, thus avoiding unnecessary emergency operation. In adults presenting with early-uncomplicated acute appendicitis, this management pathway is still uncertain and most randomized controlled trials (RCT) and meta-analysis have not been able to show significant benefit of AMS over surgery management strategy (SMS), partly due to variable treatment efficacy, high recurrence rate within a year and a lack of agreement of whom would constitute a group of EuAA.

The working hypothesis of this study is that RIPASA score as a Clinical Prediction Rule, can determine a group of patients with a diagnosis of EuAA, based on the range of scores (RIPASA score 7.5 - 11.5), who will benefit from an AMS rather than SMS, leading to improve patients' outcomes through a significant reduction in negative appendicectomy rate, shorter length of hospital stay, reduce post-operative complications and changing physician behavior in managing this group of patients to an AMS rather than SMS and ultimately financial cost savings.

The primary specific aim of this study is to compare AMS with SMS in patients with EuAA in a prospective non-inferiority RCT. Secondary specific aims are to determine the range of RIPASA score that can define a group of patients with EuAA, step 3 validation of RIPASA score as a valid CPR and improve patient outcomes in terms of reducing unnecessary negative appendicectomy rate, hospital stay and complications arising from such surgery, and ultimately financial cost savings.

DETAILED DESCRIPTION:
Introduction:

Acute appendicitis is one of the most common surgical emergencies, with a lifetime prevalence approximately 1 in 7. The incidence is 1.5-1.9 per 1000 in a male and female population with approximately 1.4 times greater in men than in women.

Despite being a common problem, acute appendicitis remains a difficult diagnosis to establish, particularly in the young, elderly and female of reproductive age. Delay in surgery may risk appendicular perforation and sepsis. Reduced diagnostic accuracy and early surgery risk significantly high negative appendicectomy rate of about 20-40%. Diagnostic accuracy can be further improved by using ultrasonography or computed tomography scan. However, these modalities are costly and may not easily be available when needed.

Clinical prediction rule (CPR) such as Alvarado score, the modified Alvarado score, and the RIPASA score have been developed to improve the diagnostic accuracy of acute appendicitis. Alvarado and Modified Alvarado scores have been reported to have very low sensitivity and specificity when applied to an Asian population with a completely different ethnic origin and diet. Thus RIPASA score was developed specifically for an Asian population and have been reported to have a significantly better sensitivity (98%) and specificity (82%) over the former two scores. Since 2009, the RIPASA score has undergone broad validation in different population settings with a different prevalence of acute appendicitis across the world and reported similarly high sensitivity and specificity.

The standard management of acute appendicitis has remained largely been unchallenged since the late 19th century, largely because of the belief that if left untreated surgically, acute uncomplicated appendicitis will progress to perforation and peritonitis with increased morbidity and mortality. Furthermore current surgical management of acute appendicitis is associated with an unacceptably high negative appendicectomy rate of about 20-40% and significant post-operative complications.

Antibiotic non-operative therapy of intra-abdominal sepsis has been accepted as mainstay therapy for a condition such as diverticulitis. Since 2009, antibiotic non-operative therapy has been increasingly proposed as an alternative strategy for early uncomplicated acute appendicitis (EuAA) and has also been reported to be safe and effective in children with acute appendicitis complicated by perforation, abscess or phlegmon formation.

However, despite multiple randomized controlled trials (RCTs) and meta-analyses, the role of antibiotics in the management of EuAA in adults remains controversial. Early RCTs have reported treatment efficacy for antibiotic non-operative management strategy (AMS) of EuAA as high as 88-91% with a recurrence rate of acute appendicitis at 13-14% at 1-year follow-up. More recent RCTs comparing AMS versus surgical management strategy (SMS) have not been able to confirm non-inferiority of AMS over SMS. These later findings were also been supported by multiple recent meta-analyses. The discrepancies in reported studies are due to a lack of agreeable definition of EuAA, which was the common recommendation by all the recent meta-analyses. The NOTA study in 2014 reported using clinical prediction rules such as Acute Inflammatory Response (AIR) score (mean score of 4.9) and Alvarado score (mean score of 5.2) to define their group with EuAA, but this was only a prospective cohort study design and the mean score used were well below the threshold for diagnosing acute appendicitis.

RIPASA Score provides a range of score from 3.0-16.5 for diagnosing acute appendicitis. RIPASA score less than 7 are considered having a low probability of acute appendicitis and RIPASA score more than 7.5 are considered high probability of acute appendicitis. Thus it may be possible to identify a group of patients with EuAA based on their RIPASA score range who may benefit from AMS.

This study-working hypothesis is that RIPASA score as a CPR can determine a group of patients with a diagnosis of EuAA, who will benefit from AMS rather than SMS. The primary specific aim of this study is to confirm the non-inferiority status of AMS over SMS in EuAA. Secondary specific aims are to determine the range of RIPASA score which can be considered as providing a firm diagnosis of EuAA which can be management with AMS rather than SMS, step 3 impact analysis of RIPASA score as a CPR, and improve patient outcomes in terms of reducing unnecessary negative appendicectomy rate, hospital stay and complications arising from such surgery, and ultimately financial cost savings.

Methodology:

Trial Design:

This study also known as RIPASA-TWO trial is designed as a single center, open-label, non-inferiority, prospective RCT to compare 2 management strategies for suspected EuAA, AMS versus SMS, using RIPASA score to identify the group of patients with EuAA and to monitor the progression of the disease and guiding surgical decision based on the participants' RIPASA score.

Population and Study Setting:

The study setting will be based at Raja Isteri Pengiran Anak Saleha (RIPAS) Hospital, a tertiary referral center. All staffs of the Department of General Surgery (GS) and Accident & Emergency (A&E) Department at RIPAS Hospital will be brief of the trial design and purpose.

Recruitment:

Patients presenting to A&E Department at RIPAS Hospital with right iliac fossa pain will be triaged and seen by the Casualty Officer. RIPASA score will be derived. Patients with RIPASA score between 7.5 to 11.5 and who satisfy the study inclusion and exclusion criteria will be referred to the on-call surgical medical officer (MO) for recruitment to RIPASA-TWO trial. Antibiotics will be withheld until patients have been seen by the surgical MO on duty and the RIPASA score is confirmed. The Surgical MO will inform and explain to the patient and family of the study and a study information sheet will be provided. Upon written signed consent to be recruited for the RIPASA-TWO trial, patients will be randomized to either arms - AMS or SMS.

Allocation concealment:

A variable block randomization sequence of 4,6 and 8 will be used to allocate participants to either AMS or SMS. A web-based program will be used and accessed via secured username and password, to obtain randomization allocation for the recruited participants. Once the randomization allocation code has been given, the surgical MO will allocate the treatment according to the randomized arm. Recruitment will be stratified to two RIPASA score range, 7.5-9.5 and 10.0-11.5.

Study Protocol:

The surgical MO/SMO will login into the randomization allocation software to acquire the randomization allocation arm and code. The patient will then be admitted to GS inpatient wards. Patients randomized to AMS arm will receive the allocated antibiotic treatment. Those randomized to SMS arm will receive the usual Departmental antibiotic policy of preoperative antibiotics prior to appendicectomy.

For patients in the AMS arm, the RIPASA score will be repeated to monitor the progression of the patient's condition after 24 hours. If RIPASA score remains stable or decreasing, the patient will continue on the allocated intravenous (iv) antibiotic treatment. If RIPASA score is increasing but remain below 11.5, the team looking after the patient can consider ordering further investigations such as ultrasound or CT scan, but patients will continue at this point on the antibiotic. If the RIPASA score increases to above 12, the surgeon can consider appendicectomy.

For patients in the AMS arm who have not cross over to surgery, they will continue with iv antibiotics for 48 hours and if symptoms improved with decreasing RIPASA score to below 7.5, the antibiotic will be changed to oral route and the patient monitored regularly. If RIPASA score goes below 5, the patient can be considered for discharge and follow-up in 1 week in the clinic with an oral antibiotic for a total of 7 days.

For patient randomized to the SMS arm, patients will undergo appendicectomy, unless their repeated RIPASA score decreases to below 7.5 or if their symptoms improved. For these patients, they will remain on iv antibiotics and will be changed to oral route after 48 hours. If RIPASA score goes below 5, the patient can be considered for discharge and follow-up in 1 week in the clinic with an oral antibiotic for a total of 7 days.

Antibiotic:

Intravenous Amikacin 15mg/kg/day divided over 3 doses for 48 hours will be the antibiotic of choice for RIPASA-TWO trial and is based on the microbial antibiotic sensitivity from pus swab taken for all appendicectomy from the previous year (2016). After 48 hours, this will be converted to oral ciprofloxacin 500mg bd for 7 days. For patients allocated to SMS arm, the Department antibiotic policy is for a preoperative antibiotic combination of intravenous Cefuroxime 1.5g TDS and 500mg metronidazole TDS.

Statistical methods:

Sample size calculation:

According to Chong et al, the reported negative appendicectomy rate based on the RIPASA score was 14.7%. Hence this 14.7% can be considered as surgical treatment failure due to an unnecessary operation and the surgical treatment efficacy is about 85.3%.

The non-inferiority margin for RIPASA-TWO trial will be set based on this surgical treatment failure rate of 14.7%. Using the FDA-approved non-inferiority margin of 50% reduction in efficacy or 50% increase in failure rate will give AMS an acceptable failure rate of 22%. Thus a treatment failure for AMS between 14-22% will be considered as confirmation of non-inferiority. A treatment failure of less than 14% will be considered as superiority. Hence based on a difference in treatment efficacy rate of 7% (22% vs 14%), with a sample size powered at 80% at 5% significance, the sample size needed to show non-inferiority is 91 in each group. Assuming a dropout rate of 25%, the total number of patients needed to be recruited is 228 patients, based on a 1:1 recruitment.

All statistical analysis will be performed using SPSS statistical program. Categorical data will be presented using frequencies and percentages. Continuous data will be presented as mean ± SD. All analysis will be conducted based on intention-to-treat principle and per-protocol analysis. Statistical analysis for categorical data will be carried out using Chi Square exact test. Differences between groups with normally distributed variables will be tested using independent sample t-test. Variables with no normal distribution will be tested using Wann-Whitney test. Non-inferiority for AMS will be tested using one-sided Wald tests with an α level of 0.05.

Duration of Study:

Based on the previous study, the recruitment of 200 consecutive patients with acute appendicitis, took over 8 months. Half of this group had RIPASA score from 7.5 to 11.5. Thus for a sample size of 228 for the RIPASA-TWO trial, the expected recruitment time is about 19 months. Hence the study will be expected to complete within 2 years.

Interim Analysis:

An interim analysis will be conducted at 2-time points. For changes to antimicrobial sensitivity, the interim analysis will be conducted at every 6 months and any changes will be discussed with the Data Safety Monitoring Board for proposed changes to the antibiotic regime. The main study interim analysis will be conducted at 1-year post recruitment to assess safety efficacy of the trial to ensure that not too many patients are developing complicated acute appendicitis in the AMS arm.

Ethical Consideration:

Ethics approval for the study has been granted by the Medical and Health Research and Ethics Committee based in RIPAS Hospital.

ELIGIBILITY:
Inclusion Criteria:

* More than 12 years of age
* High probability of early-uncomplicated acute appendicitis with confirmed RIPASA score of 7.5 to 11.5

Exclusion Criteria:

* 12 years of age or less
* RIPASA score 7 or less, or greater than 12
* Clinical diagnosis of acute complicated appendicitis with perforation or signs of generalized peritonitis.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of cases of treatment failures in each arm | 30 days
  Treatment failure for AMS is defined as cases where surgery is performed unplanned from time of randomisation up to 30 days follow up with positive histopathological confirmation of acute appendicitis (suppurative or gangrenous or perforated). Treatment failure for SMS group is defined as the unnecessary operation performed where the histopathological report is that of normal appendix, as an indicator of negative appendicectomy rate or cases who did not undergo surgery from time of randomisaton up to 30 days follow-up.

SECONDARY OUTCOMES:
Length of hospital stay | 72 to 168 hours
  Length of hospital stay from time of randomization to discharge in hours
Treatment related complications | 30 days
  30 days treatment related complications from time of randomization which will include:
  a. Antibiotic non-operative management group i. Appendiceal perforation ii. Peritonitis iii. Abscess or phlegmon formation b. Observation/Surgery i. Surgical site infection ii. Bowel obstruction secondary to bowel adhesions iii. Sepsis
Recurrence rate | 1 year
  Recurrence rate at any time of follow up > 1 month, and up to 12 months. Recurrence is defined as readmission for suspected acute appendicitis or subsequently proven to be acute appendicitis on histological specimen following surgery for AMS group after discharge. Recurrence will not be categorise as treatment failure in the AMS group since the appendix has not been surgically removed and patients in this group although at a higher rate of recurrence of about 13-14% at 1year follow up, does not represent failure of treatment for the initial episode of acute appendicitis.
Treatment cost in US dollar | 1 year
  Treatment cost in US dollar, calculated at completion of study and follow up at 1 year post randomization, which will include all radiological examinations carried out during the study period related to the condition of study.
Defining a group with RIPASA score range where AMS is most beneficial | 30 days
  Defining a group with RIPASA score range where AMS is most beneficial
Number of medical sick leave days taken | 1 year
  Number of medical sick leave days taken off work related to condition of study
Number of cases of non-compliance to RIPASA Score guidelines | 30 days
  Physician change behavior is measured through compliance rate with using the RIPASA score and adherence to RIPASA score guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Chee Fui Chong, FRCSEd, Principal Investigator — RIPAS Hospital
Locations (1):
- Raja Isteri Pengiran Anak Saleha Hospital, Bandar Seri Begawan, Daerah Brunei dan Muara, Brunei

IPD SHARING:
Plan to Share IPD: No
Written request to Ministry of Health, Brunei Darussalam via Principal Investigator for approval to share IPD.

REFERENCES:
- [Background] Stephens PL, Mazzucco JJ. Comparison of ultrasound and the Alvarado score for the diagnosis of acute appendicitis. Conn Med. 1999 Mar;63(3):137-40. PMID 10218289
- [Background] Cusheri A. The small intestine and vermiform appendix. In: In: Cuscheri A, Giles GR, Mossa AR, eds Essential Surgical Practice. 3rd ed. Oxford: Butterworth-Heinermann; p. 1297-329, 1995.
- [Background] Gilmore OJ, Browett JP, Griffin PH, Ross IK, Brodribb AJ, Cooke TJ, Higgs MJ, Williamson RC. Appendicitis and mimicking conditions. A prospective study. Lancet. 1975 Sep 6;2(7932):421-4. doi: 10.1016/s0140-6736(75)90841-7. PMID 51235
- [Background] Velanovich V, Satava R. Balancing the normal appendectomy rate with the perforated appendicitis rate: implications for quality assurance. Am Surg. 1992 Apr;58(4):264-9. PMID 1586087
- [Background] Kalan M, Talbot D, Cunliffe WJ, Rich AJ. Evaluation of the modified Alvarado score in the diagnosis of acute appendicitis: a prospective study. Ann R Coll Surg Engl. 1994 Nov;76(6):418-9. PMID 7702329
- [Background] McGinn TG, Guyatt GH, Wyer PC, Naylor CD, Stiell IG, Richardson WS. Users' guides to the medical literature: XXII: how to use articles about clinical decision rules. Evidence-Based Medicine Working Group. JAMA. 2000 Jul 5;284(1):79-84. doi: 10.1001/jama.284.1.79. PMID 10872017
- [Background] Alvarado A. A practical score for the early diagnosis of acute appendicitis. Ann Emerg Med. 1986 May;15(5):557-64. doi: 10.1016/s0196-0644(86)80993-3. PMID 3963537
- [Background] Al-Hashemy AM, Seleem MI. Appraisal of the modified Alvarado Score for acute appendicits in adults. Saudi Med J. 2004 Sep;25(9):1229-31. PMID 15448772
- [Background] Chong CF, Adi MI, Thien A, Suyoi A, Mackie AJ, Tin AS, Tripathi S, Jaman NH, Tan KK, Kok KY, Mathew VV, Paw O, Chua HB, Yapp SK. Development of the RIPASA score: a new appendicitis scoring system for the diagnosis of acute appendicitis. Singapore Med J. 2010 Mar;51(3):220-5. PMID 20428744
- [Background] Chong CF, Thien A, Mackie AJ, Tin AS, Tripathi S, Ahmad MA, et al. Evaluation of the RIPASA score: A new scoring system for the diagnosis of acute appendicitis. Brunei International Medical Journal 6:17-26, 2010. [Accessed on 2017 May 23]. Available from: http://www.bimjonline.com/PDF/Bimj%202010%20Volume%206,%20Issue%201/chong%20et%20al%20bimj2010611726OA.pdf
- [Background] Chong CF, Thien A, Mackie AJ, Tin AS, Tripathi S, Ahmad MA, Tan LT, Ang SH, Telisinghe PU. Comparison of RIPASA and Alvarado scores for the diagnosis of acute appendicitis. Singapore Med J. 2011 May;52(5):340-5. PMID 21633767
- [Background] Regar MK, Choudhary GS, Nogia C, Pipal DK, Agrawal A, Srivastava H. Comparison of Alvarado and RIPASA scoring systems in diagnosis of acute appendicitis and correlation with intraoperative and histopathological findings. International Surgery Journal 4(5):1755-1761, 2017. DOI: http://dx.doi.org/10.18203/2349-2902.isj20171634 [Accessed on 2017 May 20]. Available from: http://www.ijsurgery.com/index.php/isj/article/viewFile/1230/1159
- [Background] Malik MU, Connelly TM, Awan F, Pretorius F, Fiuza-Castineira C, El Faedy O, Balfe P. The RIPASA score is sensitive and specific for the diagnosis of acute appendicitis in a western population. Int J Colorectal Dis. 2017 Apr;32(4):491-497. doi: 10.1007/s00384-016-2713-4. Epub 2016 Dec 15. PMID 27981378
- [Background] Abd El Maksoud W, Bawahab M, Al Shehri D, Mostafa O, Ali H, Alwail A, et al. Comparison between the validity of the "Modified Alvarado" and "Raja Isteri Pengiran Anak Saleha" scores for the diagnosis of acute appendicitis. The Egyptian Journal of Surgery 36(1):52, 2017. [Accessed on 2017 May 23]. Available from: http://www.ejs.eg.net/article.asp?issn=1110-1121;year=2017;volume=36;issue=1;spage=52;epage=57;aulast=Abd
- [Background] Subramani B, Kalaichelvan L, Selvam G, Madhavan L. Comparison between RIPASA and Alvarado scoring in diagnosing acute appendicitis. Journal of Evidence Based Medicine and Healthcare 4(11):624-7, 2017. [Accessed on 2017 May 23]. Available from: http://www.jebmh.com/data_pdf/Ganganesamy%20-%20FINAL.pdf
- [Background] Rodrigues w, Sindhu S. Diagnostic Importance of Alvarado and RIPASA Score in Acute Appendicitis. International Journal of Scientific Study 4(11):57-60, 2017. [Accessed on 2017 May 23]. Available from: http://www.ijss-sn.com/uploads/2/0/1/5/20153321/volume_4_issue_11.pdf
- [Background] Anilkumar, S, Anilkumar A, Shijina, K, Unnikrishnan, G. Diagnostic Efficacy of Ripasa Scoring in Acute Appendicitis: A Tertiary Care Centre Study. Journal of Medical Science and Clinical Research 05(01):17126-30, 2017. [Accessed on 2017 May 23]. Available from: http://jmscr.igmpublication.org/v5-i1/142%20jmscr.pdf
- [Background] Singla A, Singla S, Singh M, Singla D. A comparison between modified Alvarado score and RIPASA score in the diagnosis of acute appendicitis. Updates Surg. 2016 Dec;68(4):351-355. doi: 10.1007/s13304-016-0381-0. Epub 2016 Jun 23. PMID 27338243
- [Background] Ramzanali Damani, SAA, Hussain Shah, SS, Hashami, A, Mansoori, MS. Effective diagnosis of acute appendicitis - comparison of RIPASA and Alvarado Scoring systems. Journal of Surgery Pakistan International 21(3):88-91, 2016. [Accessed on 2017 May 23]. Available from: http://www.jsp.org.pk/
- [Background] Golden SK, Harringa JB, Pickhardt PJ, Ebinger A, Svenson JE, Zhao YQ, Li Z, Westergaard RP, Ehlenbach WJ, Repplinger MD. Prospective evaluation of the ability of clinical scoring systems and physician-determined likelihood of appendicitis to obviate the need for CT. Emerg Med J. 2016 Jul;33(7):458-64. doi: 10.1136/emermed-2015-205301. Epub 2016 Mar 2. PMID 26935714
- [Background] Muduli IC, Rout BK, Mallick SN. Comparison of RIPASA AND Alvarado score in diagnosis of acute appendicitis. Journal of Evolution of Medical and Dental Sciences 5(33):1794-1798, 2016. Doi: 10.14260/jemds/2016/423. [Accessed on 2017 May 23]; Available from: https://www.jemds.com/data_pdf/Bismaya%20Kumar%20Rout.pdf
- [Background] Verma M, Vashist MG, Goyal K, Yadav P, others. Comparision of Alvarado And Ripasa Scoring Systems in Diagnosis of Acute Appendicitis. PARIPEX-Indian Journal of Research 4(8):55-57, 2016. [Accessed on 2017 May 23]. Available from: https://www.worldwidejournals.com/paripex/file.php?val=August_2015_1438856332__20.pdf
- [Background] Sinnet P, Chellappa PM, Kumar S, Ethirajulu R, Thambi S. Comparative study on the diagnostic accuracy of the RIPASA score over Alvarado score in the diagnosis of acute appendicitis. Journal of Evidence Based Medicine and Healthcare 3(80):4318-21, 2016. [Accessed on 2017 May 23]. Available from: http://www.jebmh.com/data_pdf/Peter%20Manoharan%20--%20FINAL.pdf
- [Background] Rathod S, Ali I, Bawa AS, Singh G, Mishra S, Nongmaithem M. Evaluation of Raja Isteri Pengiran Anak Saleha Appendicitis score: A new appendicitis scoring system. Medical Journal Dr. D.Y. Patil University 8(6):744, 2015. [Accessed on 2017 May 23]. Available from: http://www.mjdrdypu.org/article.asp?issn=0975-2870;year=2015;volume=8;issue=6;spage=744;epage=749;aulast=Rathod
- [Background] Khadda S, Yadav AK, Ali A, Parmar A, Sakrani JK, Beniwal H. CLINICAL STUDY TO EVALUATE THE RIPASA SCORING SYSTEM IN THE DIAGNOSIS OF ACUTE APPENDICITIS. American Journal of Advanced Medical & Surgical Research 1(2):67-73, 2015. [Accessed on 2017 Mar 27]; Available from: http://mcmed.us/downloads/1452675139(ajamsr).pdf
- [Background] Liu W, Wei Qiang J, Xun Sun R. Comparison of multislice computed tomography and clinical scores for diagnosing acute appendicitis. J Int Med Res. 2015 Jun;43(3):341-9. doi: 10.1177/0300060514564475. Epub 2015 Mar 11. PMID 25762518
- [Background] Karan M, Mukesh MK. Significance of Ripasa Scoring System in Diagnosis f Acute Appendicitis. International Journal of Healthcare Science 3(1):4-10, 2015. [Accessed on 2017 May 23]. Available from: http://www.researchpublish.com/journal/IJHS/Issue-1-April-2015-September-2015/60
- [Background] N N, Mohammed A, Shanbhag V, Ashfaque K, S A P. A Comparative Study of RIPASA Score and ALVARADO Score in the Diagnosis of Acute Appendicitis. J Clin Diagn Res. 2014 Nov;8(11):NC03-5. doi: 10.7860/JCDR/2014/9055.5170. Epub 2014 Nov 20. PMID 25584259
- [Background] Butt MQ, Chatha SS, Ghumman AQ, Farooq M. RIPASA score: a new diagnostic score for diagnosis of acute appendicitis. J Coll Physicians Surg Pak. 2014 Dec;24(12):894-7. PMID 25523723
- [Background] Alnjadat I, Abdallah B. Alvarado versus RIPASA score in diagnosing acute appendicitis. Rawal Medical Journal 38(2):147-51, 2013. [Accessed on 2017 May 23]. Available from: http://www.ejmanager.com/fulltextpdf.php?mno=28231
- [Background] Erdem H, Cetinkunar S, Das K, Reyhan E, Deger C, Aziret M, Bozkurt H, Uzun S, Sozen S, Irkorucu O. Alvarado, Eskelinen, Ohhmann and Raja Isteri Pengiran Anak Saleha Appendicitis scores for diagnosis of acute appendicitis. World J Gastroenterol. 2013 Dec 21;19(47):9057-62. doi: 10.3748/wjg.v19.i47.9057. PMID 24379631
- [Background] Reyes-García N, Zaldívar-Ramírez FR, Cruz-Martínez R, Sandoval-Martínez MD, Gutiérrez-Banda CA, Athié-Gutiérrez C. Precisión diagnóstica de la escala RIPASA para el diagnóstico de apendicitis aguda: análisis comparativo con la escala de Alvarado modificada. Cirujano General 34(2):101-6, 2012. [Accessed on 2017 May 23]. Available from: http://www.scielo.org.mx/scielo.php?script=sci_arttext&pid=S1405-00992012000200002
- [Background] Klabtawee W, Saensak W, Khetsoongnern A, Piriyasupong T. Accuracy of RIPASA and Modified RIPASA score Comparing with Alvarado Score for Diagnosis of Acute Appendicitis and Complication of Acute Appendicitis. Khon Kaen Medical Journal 35(1):38-47, 2011. [Accessed on 2017 May 23]. Available from: http://thailand.digitaljournals.org/index.php/KKMJ/article/view/7108
- [Background] Resende F, Almeida AB, Costa Maia J, Bessa Melo R. Challenges in uncomplicated acute appendicitis. Journal of Acute Disease 5(2):109-13, 2016. [Accessed on 2017 May 23]. Available from: http://ac.els-cdn.com/S2221618916000056/1-s2.0-S2221618916000056-main.pdf?_tid=9b43f614-3f7a-11e7-abbd-00000aab0f27&acdnat=1495518328_a700b453b724f58fc38c6f99b72aeadd
- [Background] Di Saverio S, Sibilio A, Giorgini E, Biscardi A, Villani S, Coccolini F, Smerieri N, Pisano M, Ansaloni L, Sartelli M, Catena F, Tugnoli G. The NOTA Study (Non Operative Treatment for Acute Appendicitis): prospective study on the efficacy and safety of antibiotics (amoxicillin and clavulanic acid) for treating patients with right lower quadrant abdominal pain and long-term follow-up of conservatively treated suspected appendicitis. Ann Surg. 2014 Jul;260(1):109-17. doi: 10.1097/SLA.0000000000000560. PMID 24646528
- [Background] Antibiotic therapy for acute appendicitis in adults. Fewer immediate complications than with surgery, but more subsequent failures. Prescrire Int. 2014 Jun;23(150):158-60. PMID 25121154
- [Background] Styrud J, Eriksson S, Nilsson I, Ahlberg G, Haapaniemi S, Neovius G, Rex L, Badume I, Granstrom L. Appendectomy versus antibiotic treatment in acute appendicitis. a prospective multicenter randomized controlled trial. World J Surg. 2006 Jun;30(6):1033-7. doi: 10.1007/s00268-005-0304-6. PMID 16736333
- [Background] Hansson J, Korner U, Khorram-Manesh A, Solberg A, Lundholm K. Randomized clinical trial of antibiotic therapy versus appendicectomy as primary treatment of acute appendicitis in unselected patients. Br J Surg. 2009 May;96(5):473-81. doi: 10.1002/bjs.6482. PMID 19358184
- [Background] Vons C, Barry C, Maitre S, Pautrat K, Leconte M, Costaglioli B, Karoui M, Alves A, Dousset B, Valleur P, Falissard B, Franco D. Amoxicillin plus clavulanic acid versus appendicectomy for treatment of acute uncomplicated appendicitis: an open-label, non-inferiority, randomised controlled trial. Lancet. 2011 May 7;377(9777):1573-9. doi: 10.1016/S0140-6736(11)60410-8. PMID 21550483
- [Background] Varadhan KK, Humes DJ, Neal KR, Lobo DN. Antibiotic therapy versus appendectomy for acute appendicitis: a meta-analysis. World J Surg. 2010 Feb;34(2):199-209. doi: 10.1007/s00268-009-0343-5. PMID 20041249
- [Background] Wilms IM, de Hoog DE, de Visser DC, Janzing HM. Appendectomy versus antibiotic treatment for acute appendicitis. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD008359. doi: 10.1002/14651858.CD008359.pub2. PMID 22071846
- [Background] Harnoss JC, Zelienka I, Probst P, Grummich K, Muller-Lantzsch C, Harnoss JM, Ulrich A, Buchler MW, Diener MK. Antibiotics Versus Surgical Therapy for Uncomplicated Appendicitis: Systematic Review and Meta-analysis of Controlled Trials (PROSPERO 2015: CRD42015016882). Ann Surg. 2017 May;265(5):889-900. doi: 10.1097/SLA.0000000000002039. PMID 27759621
- [Background] Fitzmaurice GJ, McWilliams B, Hurreiz H, Epanomeritakis E. Antibiotics versus appendectomy in the management of acute appendicitis: a review of the current evidence. Can J Surg. 2011 Oct;54(5):307-14. doi: 10.1503/cjs.006610. PMID 21651835
- [Background] Podda M, Cillara N, Di Saverio S, Lai A, Feroci F, Luridiana G, Agresta F, Vettoretto N; ACOI (Italian Society of Hospital Surgeons) Study Group on Acute Appendicitis. Antibiotics-first strategy for uncomplicated acute appendicitis in adults is associated with increased rates of peritonitis at surgery. A systematic review with meta-analysis of randomized controlled trials comparing appendectomy and non-operative management with antibiotics. Surgeon. 2017 Oct;15(5):303-314. doi: 10.1016/j.surge.2017.02.001. Epub 2017 Mar 9. PMID 28284517
- [Background] GUIDANCE D. Preparation of Food Contact Notifications for Food Contact Substances in Contact with Infant Formula and/or Human Milk: Guidance for Industry. Cent Food Saf Appl Nutr [Internet]. 2016 [Accessed on 2017 Apr 18]; Available from: https://www.fda.gov/downloads/Food/GuidanceRegulation/GuidanceDocumentsRegulatoryInformation/UCM528255.pdf
- [Background] Sealed Envelope | Power calculator for binary outcome non-inferiority trial [Internet]. [Accessed on 2017 Apr 24]. Available from: https://www.sealedenvelope.com/power/binary-noninferior/